CLINICAL TRIAL: NCT03245580
Title: Comparison of 2 Techniques Using EUS Guided Liver Biopsies Via 19g CORE Biopsy Needle to Obtain Optimal Core Liver Biopsies in Benign Disease
Brief Title: Benign Liver Optimal Core Study (Tissue Acquisition Comparison in Benign Liver Disease)
Acronym: BLOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkview Health (Other)
Responsible Party: Principal Investigator, Neil Sharma, M.D., President, Parkview Cancer Institute;Director Advanced Interventional Endoscopy & Endoscopic Oncology, Parkview Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRC17-0714
Record Dates: First submitted 2017-07-17; First posted 2017-08-10 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: prospective, randomized, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1 -modified wet suction (Other): Intervention:Procedure Core Liver Biopsy Technique: Modified Wet Suction
  Interventions: Diagnostic Test: Core Liver Biopsy
- Arm 2- Slow Pull (Other): Intervention: Procedure Core Liver Biopsy Technique: Slow Pull
  Interventions: Diagnostic Test: Core Liver Biopsy

INTERVENTIONS:
Diagnostic Test: Core Liver Biopsy — Diagnostic EUS examination followed by liver biopsy to obtain core sample in benign liver disease.

SUMMARY:
The primary purpose of this prospective, randomized, multicenter study is to evaluate and compare the amount and quality of tissue samples yielded in a liver biopsy comparing 2 different techniques of EUS guided CORE liver biopsy for benign disease. The two techniques: "modified Wet suction" and "Slow pull" technique of collecting tissue from a liver biopsy via Endoscopic Ultrasound (EUS).

DETAILED DESCRIPTION:
Each subject will have a biopsy performed via one of 2 different techniques: "modified wet suction", or "slow pull" technique. A randomization process will determine which technique. Each subject shall undergo 2 passes (2 cores of tissue will be obtained - ideally from the right and left lobe of the liver.

Quality of tissue obtained via the 2 different techniques will be evaluated by number of fragments, length of specimens and number of tracts observed by the local pathologist and compared between the tissues obtained from the two techniques. .

ELIGIBILITY:
Inclusion Criteria:

* Subjects that plan to undergo a liver biopsy via EUS to confirm possible underlying liver disease or to determine stage, grade and presence of fibrosis for suspected benign etiology.
* History of abnormal LFTs
* Documented history of chronic liver disease
* Question of underlying liver disease as cause of abnormal imaging or symptoms which may be attributed to liver disorder
* Fatty liver disease
* Subjects 18 years of age or older
* Subject must be able to hold anticoagulants as per institutional standard of care
* Subjects must be deemed physically able to undergo anesthesia. This includes either Monitored Anesthesia Care (MAC) or general anesthesia.
* Subjects (or the subjects Legally Authorized Representative [LAR]) that have agreed to participate in the study and have signed Informed Consent
* Women of child bearing potential who are not pregnant as proven by a negative pregnancy test may be included.

Exclusion Criteria

* Subjects that are unable to tolerate anesthesia for the procedure
* Subjects 17 or under
* Subjects whose anticoagulants cannot be held
* Subjects who cannot have or refuse EUS guided procedure
* Subjects who are pregnant
* INR >1.5
* Platelets 50,000 or less
* Subjects requiring control of bleeding on initial upper endoscopy
* Subjects requiring endoscopic mucosal resection
* Subjects with large volume ascites
* Subjects requiring pancreatic biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil R Sharma, MD, Principal Investigator — parkview cancer institute
Locations (7):
- United States (7):
  - University South Alabama, Mobile, Alabama
  - Santa CLara Valley Medical Center, San Jose, California
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University, Indianapolis, Indiana
  - Oschner Health System, New Orleans, Louisiana
  - Geisinger Medical Center, Danville, Pennsylvania
  - Baylor Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 -Modified Wet Suction | Arm 2- Slow Pull
Started | 75 | 78
Completed | 75 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 -Modified Wet Suction | Arm 2- Slow Pull | Total
Number analyzed (Participants) | 75 | 78 | 153
Age, Continuous [Median (Full Range); unit: years] | 55.1 [46.8 to 63.3] | 56.6 [48.4 to 64.1] | 55.85 [46.8 to 64.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 44 | 104
  Male | 15 | 34 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 70 | 71 | 141
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 65 | 66 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 75 | 76 | 153
Hypertension [Count of Participants; unit: Participants] | 37 | 39 | 76
Diabetic [Count of Participants; unit: Participants] | 27 | 23 | 50
Anticoagulants/Antiplatelet Therapy [Count of Participants; unit: Participants] | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Pathological Yield Fragmentation
Description: To determine if there is a significant difference in pathological yield as determined by fragmentation of portal tracts of the biopsy sample between a "modified wet suction," and "slow pull" techniques in obtaining CORE of histologic tissue. Pathological yield will be measured by assessment of portal tracts fragmentation by designated pathologists with experience in liver biopsy specimens.
Time Frame: At day 7 post biopsy
Measure: Mean (Full Range); unit: mm
Units Other Than Participants: Total number liver biopsy specimens
Arm/Group | Arm 1 -Modified Wet Suction | Arm 2- Slow Pull
Number analyzed (Participants) | 75 | 78
Number analyzed (Total number liver biopsy specimens) | 150 | 154
mm
  Length of Longest Fragment- Left Lobe | 14 [11 to 20] | 11 [6 to 15]
  Length of Longest Fragment- Right Lobe | 13 [9 to 19] | 10 [8 to 15]

2. Primary Outcome: Pathological Yield Length
Description: To determine if there is a significant difference in pathological yield as determined by length of portal tracts of the biopsy sample between a "modified wet suction," and "slow pull" techniques in obtaining CORE of histologic tissue. Length of portal tracts will be measured in mm by designated pathologists with experience in liver biopsy assessment techniques.
Time Frame: At time of completion of pathology report
Measure: Mean (Full Range); unit: mm
Units Other Than Participants: Number of liver biopsy specimens
Arm/Group | Arm 1 -Modified Wet Suction | Arm 2- Slow Pull
Number analyzed (Participants) | 75 | 78
Number analyzed (Number of liver biopsy specimens) | 147 | 151
mm
  Total Length of Fragments - Left Lobe | 46.5 [31 to 71] | 34.5 [17 to 42]
  Total Length of Fragments-Right Lobe | 38 [22 to 60] | 28 [17 to 40]

3. Primary Outcome: Pathological Yield Quantity
Description: To determine if there is a significant difference in pathological yield as determined by number of portal tracts of the biopsy sample between a "modified wet suction," and "slow pull" techniques in obtaining CORE of histologic tissue. The number of portal tracts will be assesses and tallied by designated pathologists with experience in the assessment of liver biopsies.
Time Frame: At time of completion of pathology report
Measure: Mean (Full Range); unit: Number of portal tracts
Units Other Than Participants: Number of liver biopsy specimens
Arm/Group | Arm 1 -Modified Wet Suction | Arm 2- Slow Pull
Number analyzed (Participants) | 75 | 78
Number analyzed (Number of liver biopsy specimens) | 150 | 154
Number of portal tracts
  Total Number of Portal Tracts Left Lobe | 16 [12 to 24.5] | 11.5 [6.5 to 18.5]
  Total Number of Portal Tracts Right Lobe | 14 [10 to 18] | 12 [7 to 17]

4. Secondary Outcome: Complications
Description: Tracking any complications that may be associated with each technique. Complications will be assessed and tracked following CTCAE V4.
Time Frame: Complications occurring at time of consent, at procedure time and at day 7 post procedure
Measure: Number; unit: Number of Adverse Events
Arm/Group | Arm 1 -Modified Wet Suction | Arm 2- Slow Pull
Number analyzed (Participants) | 75 | 78
Number of Adverse Events
  Minor Adverse Events Grade 1 | 10 | 4
  Minor Adverse Events Grade 2 | 1 | 4
  Minor Adverse Events Grade 3 | 2 | 2
  Serious Adverse Events Grade 1 | 7 | 2

ADVERSE EVENTS:
Time Frame: Data collected for one week following procedure
Arm/Group | Arm 1 -Modified Wet Suction | Arm 2- Slow Pull
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/78
Serious Adverse Events (participants affected / at risk) | 7/75 | 2/78
Other Adverse Events (participants affected / at risk) | 13/75 | 10/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 -Modified Wet Suction (N=75) | Arm 2- Slow Pull (N=78)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Intraabdominal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 -Modified Wet Suction (N=75) | Arm 2- Slow Pull (N=78)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank Pain (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Fall from bed
Bronchial Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT03245580/Prot_SAP_000.pdf